CLINICAL TRIAL: NCT00001152
Title: Pigment Dispersion Syndrome With and Without Glaucoma
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 760189; 76-EI-0189
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1998-05

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension
Keywords: Aqueous Humor Dynamics; Glaucoma; Ocular Hypertension; Pigment Dispersion Syndrome; Primary Open Angle Glaucoma; Pseudo-Exfoliation of the Lens Capsule
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma-Related Pigment Dispersion Syndrome

SUMMARY:
To compare patients having PDS without and with OH or GL by documenting and following the clinical features and course of their disease and evaluating the patient's performance on a variety of diagnostic tests.

DETAILED DESCRIPTION:
Pigment dispersion syndrome (PDS) is not an uncommon ocular condition and is frequently associated with myopia. There is loss of pigment from the posterior iris, seen clinically in most cases as iris transillumination with pigment deposited on the corneal endothelium, iris surface and on the angle structures overlying Schlemm's canal. In a subset of patients ocular hypertension or glaucoma may develop.

Ocular hypertension is defined as 3 separate measurements of the intraocular pressure greater than 22 mm/Hg in the absence of visual field loss. Glaucoma is defined as the presence of a characteristic field defect (Bjerrum scotoma, nasal step or arcuate scotomas) with intraocular pressures greater than 22 mm/Hg measured sometime during a diurnal curve testing.

The etiology of this condition is not known. Hypotheses include developmental abnormalities of the iris dilator muscle or mechanical rubbing of zonules against the iris, resulting in pigment dispersion in the anterior chamber and pressure elevation. PDS is then viewed as a variant of primary open-angle glaucoma or may be secondary to pigment deposited in the angle structures with secondary damage to the trabecular meshwork. A hereditary component does appear to play a role in the PDS syndrome and may also predispose to the development of glaucoma.

The purpose of this study is to evaluate and determine the risk factors that differentiate patients with PDS, PDS+OH, or PDS+GL by documenting the ophthalmic findings and following their clinical course. In order to do this, diagnostic tests including intraocular pressure and visual fields will be performed. This data may make it possible to determine the risk of patients having PDS of developing OH, GL or other possibly associated findings such as retinal detachment or cataract. In addition, patients with "pigmentary glaucoma (PG)" will be compared to those with the known characteristics of primary open-angle glaucoma (POAG) to determine whether PG is different than or a variant of POAG. When possible, family members will be examined to investigate the inheritance pattern of this syndrome and its relationship to POAG.

ELIGIBILITY:
Entrance into the study will depend upon clinical evidence of black pigment deposition on trabecular meshwork at the site of Schlemm's canal and at least one of the following: Kruckenberg spindle, pigment deposition on iris surface, or mid-stromal iris transillumination.

No patients with other ocular disease or disorders (uveitis, trauma, pseudoexfoliation, ICE syndrome, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175
Dates: Start 1976-06; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kupfer C, Kuwabara T, Kaiser-Kupfer M. The histopathology of pigmentary dispersion syndrome with glaucoma. Am J Ophthalmol. 1975 Nov;80(5):857-62. doi: 10.1016/0002-9394(75)90283-4. PMID 1190279
- [Background] Campbell DG. Pigmentary dispersion and glaucoma. A new theory. Arch Ophthalmol. 1979 Sep;97(9):1667-72. doi: 10.1001/archopht.1979.01020020235011. PMID 475638
- [Background] Andersen JS, Pralea AM, DelBono EA, Haines JL, Gorin MB, Schuman JS, Mattox CG, Wiggs JL. A gene responsible for the pigment dispersion syndrome maps to chromosome 7q35-q36. Arch Ophthalmol. 1997 Mar;115(3):384-8. doi: 10.1001/archopht.1997.01100150386012. PMID 9076212